CLINICAL TRIAL: NCT05635448
Title: Better Together Physician Coaching: Addressing Burnout Amongst Clinicians
Brief Title: Better Together Physician Coaching to Mitigate Burnout Amongst Clinicians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 22-2158
Record Dates: First submitted 2022-11-21; First posted 2022-12-02 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Burnout, Professional; Self Compassion; Flourishing; Imposter Syndrome; Moral Injury; Loneliness
MeSH Terms: conditions — Burnout, Professional; imposter syndrome; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial. All enrolled participants will complete the pretest baseline survey. After baseline data collection is completed, the participants will be randomized into either a control or intervention group. This randomized controlled trial study design will offer the BT coaching to the intervention group for the duration of 4-months (February 1st 2023- May 31st 2023) and to the control group for the duration of 4-months (September 1st 2023 - December 31st 2023).
  At two different timepoints, all participants will be offered surveys containing the following validated indices: burnout, imposter syndrome, self-compassion, moral injury, discrimination, and flourishing. All participants will be offered the survey at baseline- January 2023 (T0), post intervention- May 2023 (T1).
Who Masked: Outcomes Assessor
Masking Description: Data will be de-identified prior to analysis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Will be offered the BT coaching intervention over 4-months (February 1st 2023- May 31st 2023).
  Interventions: Behavioral: Better Together Physician Coaching Program
- Waitlist control (Placebo Comparator): Will be offered the coaching intervention following 4-month waitlist control (September 1st 2023 - December 31st 2023).
  Interventions: Behavioral: No intervention - waitlist control

INTERVENTIONS:
Behavioral: Better Together Physician Coaching Program — thought-based coaching. This type of coaching focuses on thoughts and beliefs. It combines a cognitive behavioral therapy (CBT) model with mindfulness-based awareness and integrates theories of acceptance and commitment therapy (ACT), nonattachment, and radical questioning from Socratic and Greek philosophies. BT delivers a robust coaching experience via a 4-month web-based, group-coaching model. This novel program allows residents to participate as actively as they are inclined and able, offering flexibility via multiple modalities of coaching: twice weekly group coaching calls, unlimited anonymous written coaching, and weekly self-study modules that are housed on a secure members-only website.
  Arms: Intervention
Behavioral: No intervention - waitlist control — No intervention - waitlist control
  Arms: Waitlist control

SUMMARY:
Better Together Physician Coaching ("Better Together", or "BT"), a 4-month, web-based positive psychology multimodal coaching program was built to decrease burnout in medical trainees. Here, the investigators seek to understand it's efficacy in University of Colorado School of Medicine (CU SOM) clinicians

Aim 1: Implement Better Together in University of Colorado School of Medicine clinicians Aim 2: Assess outcomes: primary: reduce burnout as measured by the Maslach Burnout Index (goal: 10% relative improvement), and secondary: self-compassion, imposter syndrome, flourishing, loneliness, and moral injury.

Aim 3: Advance the field of coaching for clinicians through innovation and dissemination of evidence-based approaches to clinician wellbeing.

DETAILED DESCRIPTION:
Burnout refers to feelings of exhaustion, negativism, and reduced personal efficacy resulting from chronic workplace stress. In healthcare, burnout leads to increased medical errors, poorer patient care and negatively affects professional development and retention. Burnout is a growing problem that begins early in medical training. Professional coaching is a metacognition tool with a sustainable positive effect on physician well-being but typically relies on expensive consultants or time-consuming faculty development, often making it infeasible for medical training programs to offer. To overcome this barrier, the investigators created Better Together Physician Coaching (BT) a 4-month coaching program for at the University of Colorado (CU). BT includes regular online group-coaching, written coaching, and weekly self-study modules delivered by physician life coaches (Co-PIs). In 2021, the investigators studied BT in a group of female-identifying resident trainees at CU and found that the program significantly improved burnout, imposter syndrome, and self-compassion. This finding supports previous data that life coaching is effective for physicians and physicians in training. The investigators initially focused on women since burnout affects women to a greater degree than their male counterparts, and may have long-lasting consequences on their careers, contributing to a "leaky pipeline" effect. The pilot randomized controlled trial (RCT) of 101 BT women participants demonstrated a statistically significant improvement in burnout, self-compassion, and imposter syndrome in the intervention group.

The investigators now seek to understand if the coaching program is also effective in clinicians of all gender identities.

The hypothesis is that Better Together Physician Coaching ("Better Together", or "BT"), a 4-month, web-based positive psychology multimodal coaching program will result in decreased burnout in University of Colorado School of Medicine (CU SOM) clinicians.

Aim 1: Implement Better Together in CU SOM clinicians Aim 2: Assess outcomes: primary: reduce burnout as measured by the Maslach Burnout Index (goal: 10% relative improvement), and secondary: self-compassion, imposter syndrome, flourishing, loneliness, and moral injury.

Aim 3: Advance the field of coaching for clinicians through innovation and dissemination of evidence-based approaches to clinician wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* University of Colorado School of Medicine (CU SOM) clinicians AND
* Faculty

Exclusion Criteria:

* Non-CU SOM clinicians, non-faculty

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Burnout as defined by the Maslach Burnout Inventory (MBI): Change from pre to post test | pretest will occur prior to the intervention and posttest will occur after the 4-month intervention.
  The Maslach burnout inventory (MBI) is a 22-item measurement of worker burnout which assesses emotional exhaustion (EE), depersonalization (DP), and personal fulfillment (PF) domains. Possible scores range from 0-6 on a Likert scale for each item. Scores of EE ≥ 27 points, DP ≥ 10, and PF <33 would indicate a high degree of burnout. Scores of EE≤18 points, DP≤5 points, and PF≥40 points would indicate a low degree of burnout.

SECONDARY OUTCOMES:
Self-Compassion as defined by Neff's Self Compassion Score Short Form (SCS-SF): Change from pre to post test | pretest will occur prior to the intervention and posttest will occur after the 4-month intervention
  Neff's Self Compassion Score Short Form (SCS-SF) is a 12-item measurement of self-compassion. Possible scores range from 0-6 on a Likert scale for each item, where the higher scale scores indicate greater self-compassion. Scores of 1.0- 2.49 are considered to be low, between 2.5-3.5 to be moderate, and 3.51-5.0 to be high.
Moral Injury as defined by the Moral Injury Symptom Scale for Health Professions (MISS-HP): Change from pre to post test | pretest will occur prior to the intervention and posttest will occur after the 4-month intervention
  Moral Injury Symptom Scale for Health Professions (MISS-HP) is a 10-item measurement of moral injury. Possible scores range from 0-5 on a Likert scale for each item, where the higher scale scores indicate greater moral injury. Scores >35(on a possible score range of 10 to 100) are considered high for moral injury symptoms causing moderate to extreme problems with family, social, and occupational functioning.
Imposter Syndrome as defined by Young's Imposter Syndrome Symptoms Scale (YISS): Change from pre to post test | pretest will occur prior to the intervention and posttest will occur after the 4-month intervention
  Young's Imposter Syndrome Symptoms Scale (YISS) is a 8-item measurement of imposter syndrome. Scoring is yes/no where a score of >5/8 is felt to be positive for imposter syndrome.
Flourishing as defined by the Secure Flourish Index (SFI): Change from pre to post test | pretest will occur prior to the intervention and posttest will occur after the 4-month intervention
  The Secure Flourish Index (SFI) is a 12 item measurement of flourishing at work and includes the domains of (D1) happiness and life satisfaction; (D2) physical and mental health; (D3) meaning and purpose; (D4) character and virtue; and (D5) close social relationships plus 2 questions on having adequate stability as well as material and financial resources so that flourishing is likely to continue. Scores range from a low of 0 to a high of 120, though the secure flourishing scores are often reported as averages of the questions (rather than sums) so that all scores are on a scale of 0-10.
Loneliness as defined by the UCLA 3-item Loneliness Scale: Change from pre to post test | pretest will occur prior to the intervention and posttest will occur after the 4-month intervention
  The UCLA 3-item Loneliness Scale measures feelings of loneliness. It is a shortened version of the 20-item Revised UCLA Loneliness Scale. Possible scores range from 1-3 on a Likert scale for each item with 1 = Hardly ever; 2 = Some of the time; 3 = Often. The three items are summed to give a total score between 3 to 9 with higher scores indicating a higher degree of loneliness.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado School of Medicine, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Villwock JA, Sobin LB, Koester LA, Harris TM. Impostor syndrome and burnout among American medical students: a pilot study. Int J Med Educ. 2016 Oct 31;7:364-369. doi: 10.5116/ijme.5801.eac4. PMID 27802178
- [Background] Mantri S, Lawson JM, Wang Z, Koenig HG. Identifying Moral Injury in Healthcare Professionals: The Moral Injury Symptom Scale-HP. J Relig Health. 2020 Oct;59(5):2323-2340. doi: 10.1007/s10943-020-01065-w. PMID 32681398
- [Background] Kelly-Hedrick M, Rodriguez MM, Ruble AE, Wright SM, Chisolm MS. Measuring Flourishing Among Internal Medicine and Psychiatry Residents. J Grad Med Educ. 2020 Jun;12(3):312-319. doi: 10.4300/JGME-D-19-00793.1. PMID 32595851
- [Background] Fainstad T, Mann A, Suresh K, Shah P, Dieujuste N, Thurmon K, Jones CD. Effect of a Novel Online Group-Coaching Program to Reduce Burnout in Female Resident Physicians: A Randomized Clinical Trial. JAMA Netw Open. 2022 May 2;5(5):e2210752. doi: 10.1001/jamanetworkopen.2022.10752. PMID 35522281
- [Background] Maslach, C., Jackson, S. E., & Leiter, M. P. (1997). Maslach Burnout Inventory: Third edition. In C. P. Zalaquett & R. J. Wood (Eds.), Evaluating stress: A book of resources (pp. 191-218). Scarecrow Education.
- [Background] Neff KD. Self-Compassion Scale. PsycTESTS Dataset. 2012. doi:10.1037/t10178-000
- [Background] Hughes ME, Waite LJ, Hawkley LC, Cacioppo JT. A Short Scale for Measuring Loneliness in Large Surveys: Results From Two Population-Based Studies. Res Aging. 2004;26(6):655-672. doi: 10.1177/0164027504268574. PMID 18504506
- [Derived] Fainstad T, Rodriguez C, Kreisel C, Caragol J, Thibodeau PS, Kostiuk M, Mann A. Impact of an Online Group-Coaching Program on Ambulatory Faculty Physician Well-Being: A Randomized Trial. J Am Board Fam Med. 2025 Mar 21;37(6):1055-1071. doi: 10.3122/jabfm.2024.240022R1. PMID 39725465